CLINICAL TRIAL: NCT00297739
Title: Risperidone Augmentation for Treatment-Resistant Aggression in ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Armenteros, Jorge L., M.D., P.A. (Individual)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIS-ATT-401
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2006-03-16 (Estimated); Status verified 2006-03

CONDITIONS: Aggression
Keywords: Aggression; ADHD; Antipsychotic
MeSH Terms: conditions — Aggression; Attention Deficit Disorder with Hyperactivity | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
Primary objectives:

1. To assess the short-term efficacy of risperidone augmentation for treatment-resistant aggression in children with ADHD.
2. To assess the short-term safety and tolerability of risperidone augmentation in the same group of subjects.

DETAILED DESCRIPTION:
Methods and Procedures:

Study Design

The study will be a double-blind placebo-controlled trial of risperidone as an augmenting agent in 40 children, 7-12 years of age, with ADHD. All subjects would have been treated first with a stimulant medication as a single agent, but continue to present impulsive aggression. The active phase of treatment will be four weeks long, during which risperidone or placebo will be added to a constant dose of stimulant medication. The study will include a four weeks continuation phase where placebo nonresponders will have the opportunity to receive risperidone on an open basis.

Subject recruitment

Special time and effort will be devoted to subject recruitment since we recognize that it is crucial to the study. Our primary recruitment sites are the Child and Adolescent Psychiatry (CAP) outpatient clinic, the psychiatry crisis unit, and the child and adolescent psychiatry inpatient unit. Clinical staff will identify and refer to the research team potential candidates for the study. Community referrals will be sought after by means of professional liaisons and academic presentations at local psychiatric facilities. Possible subjects will then be scheduled for a full evaluation after telephone screening for inclusion and exclusion criteria. Recruitment will be continuous until the total number of proposed subjects (N=40), complete the study.

Inclusion criteria

1. Boys and girls ages 7 to 12 years, inclusive
2. Medical/neurological clearance
3. Meets DSM-IV diagnosis of ADHD
4. Treatment with a stimulant medication during the last three weeks
5. Failure to respond to stimulant medication as documented by:

   1. Three acts of aggression in the past week, two of which must be acts of physical aggression against other people, objects, or self
   2. Aggression Questionnaire (AQ) Predatory-Affective index score of 0 or below. This indicates primarily an affective or impulsive subtype of aggression
   3. Minimum CGI scale rating of 4 (moderately ill)
6. IQ > 75

Exclusion criteria

1. Major medical problems such as cardiac, renal, thyroid diseases, and seizure disorder
2. History of alcohol or substance abuse within the last 4 weeks
3. Previous adequate treatment with risperidone (2 mg/day for at least 4 weeks)
4. Acutely suicidal or homicidal
5. Unable to sign informed consent

Assessment Instruments and Scales

1. Aggression

   Understanding an aggressive episode is clearly complicated by the need to numerically quantify it. Being a low frequency behavior, aggression presents a challenge to the systematic assessment required in a research study. We will employ the Children's Aggression Scale, Parent (CAS-P) and Teacher (CAS-T) versions (Halperin et al., 2002) to measure retrospectively the frequency and severity of four categories of aggression: (1) verbal aggression, (2) aggression against objects and animals, (3) provoked physical aggression, and (4) initiated physical aggression. Responders complete a Likert scale to evaluate the frequency of an act. A distinction is made between aggressive acts directed toward persons who live in the home and those who do not, and also between acts directed toward peers and those directed towards adults. The frequency of aggressive events is multiplied by its designated severity weight factor and then summed to yield a total score. We modified the instrument so that only the occurrence of impulsive aggressive events over the previous one-week period is rated (see Appendix). These "event" types of variables fall in the category of "impulsive aggression" as defined above. Parents/guardians and teachers will be the respondents for this scale.

   Vitiello and associates (1990, 1997) studied aggressive behaviors in children and adolescents and developed the Aggression Questionnaire (AQ) to classify aggression into "predatory" and "affective" subtypes. Subsequently, Malone et al., (1998) modified the instrument by making it a parent interview and increasing the range of scoring. The modified version, which will be used in this study, is a 16-item scale consisting of eight items that assess predatory aggression and eight items that assess affective aggression. Items are scored as not true (0), partly true (1), or very true (2). Predatory and affective scores are obtained by adding the corresponding items with a possible range from 0 to 16. The Predatory-Affective index is calculated by subtracting the affective score from the predatory score. Higher index scores indicate a predominantly predatory type of aggression while lower scores indicate primarily an affective subtype. This affective aggression is viewed as an overreaction to a minor provocation often accompanied by disinhibition and behavioral dyscontrol, characteristically impulsive. The AQ differentiated responders from nonresponders to lithium treatment in a group of aggressive conduct-disordered children (Malone et al., 1998).
2. ADHD Symptoms

The Continuous Performance Test (CPT; Conners, 1995) consists of a series of letters presented on a computer screen in rapid succession. The subject is required to press a key whenever a target stimulus is presented, and to refrain from pressing the key when the nontarget stimulus is presented. The CPT generates separate measures of inattention and impulsivity. The impulsivity score is derived from a combination of commission errors and hit reaction times. T-scores of 60 or above on commission errors and hit reaction times will be considered as an indication of impulsivity.

The ADHD Index (Conners, 1997) - Because of its brevity (12 items) and excellent psychometric properties, this index is well suited for repeated measures in clinical drug trials. The ADHD Index will help us understand if the effect of risperidone treatment on impulsive aggression is independent of any effect it may have on ADHD symptomatology.

Initial visit

The initial visit will take place at the CAP outpatient clinic where the rest of the study will be conducted. The study will be fully explained and a written informed consent will be obtained from the parent(s) while an assent from will be obtained from the subject. Parent(s) and subject will undergo the following assessments:

1. Parent/Staff:

   1. Structured psychiatric interview employing the computerized Diagnostic Interview Schedule for Children IV (Generic C-DISC 4; Shaffer et al., 2000) - This is a comprehensive, structured interview that covers 36 mental health disorders for children and adolescents, using DSM-IV criteria. Extensive reliability data on this instrument are available. The instrument produces a series of reports including a diagnostic report that indicates endorsed symptoms, criteria, and diagnoses. Comorbidity in the sample will be clearly identified. The parent version is suitable for caretakers of 6 to 17 year olds. Raters will be required to participate in a two-day training session by a Columbia DISC trainer.
   2. Complete social history and review of environmental stressors
   3. Medical review of systems
   4. CAS-P, ADHD index, and AQ
2. Subject:

   1. Structured psychiatric interview employing the Generic C-DISC 4. The youth version is suitable for children aged 9 to 17 years. The parent and youth interviews will be performed in parallel except for children ages 7 and 8 years for which only the parent interview is valid.
   2. Continuous Performance Test
   3. Kaufman Brief Intelligence Test (K-BIT; Kaufman and Kaufman 1990) - The K-BIT is a brief, individually administered measure of verbal and nonverbal intelligence. While it is not intended to substitute for a comprehensive measure of intelligence, it is adequate for our screening purposes. The K-BIT IQ composite score was correlated .80 with the WISC-R full scale IQ
   4. Clinical Global Impressions (CGI) - A four-item scale widely used in clinical drug trials, involving both adult and pediatric patients.
   5. Laboratory studies will include complete blood cell count (CBC) and differential, electrolytes, thyroid and kidney function tests. These will be repeated at endpoint.
   6. Urine analysis for toxicology and pregnancy (females)
3. Teacher:

The teacher will be given the Children's Aggression Scale-Teacher Version (CAS-T) (Halperin et al., 2002) to evaluate the frequency and severity of aggressive acts, as distinct from oppositional and defiant behaviors. In addition, the teacher will be given the ADHD index. The teacher who best knows the patient will complete both scales.

The research team will discuss all information collected to arrive at a preliminary consensus diagnosis. After reviewing inclusion and exclusion criteria, subjects who are eligible will be invited to participate in the study.

Phase I

This phase will last 4 weeks. Subjects that meet inclusion criteria will be randomized to receive study medication (risperidone or placebo) as augmenting treatment to stimulant medication. The dose of the stimulant will remain constant during this phase. Janssen Pharmaceutica will supply risperidone 0.5 mg and identical placebos. All research staff and subjects will be blind as to the study medication to be administered. The dose of the study medication will be started at 0.5 mg/day. The dose for each child will be individually regulated until optimum efficacy or until the side effects become unacceptable. The guiding principle will be to achieve control of symptoms with the lowest possible dose in order to minimize undue side effects. The medication dose can be gradually increased by 0.5mg weekly to a maximum of 2 mg/day. Dose reduction for adverse events may occur at any time and be made in any multiple of 0.5 mg as deemed clinically necessary. No other concomitant medication will be permitted. Subjects will attend the research clinic on a weekly basis for behavioral assessments and medication distribution.

At the end of Phase I, the blind will be broken on every subject and the study medication will be identified. Subjects that received placebo and continue to present aggressive behaviors, as defined by inclusion criteria, will be eligible to continue to Phase II. All other subjects will be treated as clinically indicated.

Phase II

This phase will last 4 weeks. Subjects that received placebo during Phase I and continue to present aggressive behaviors will receive risperidone on an open basis. All visits, dosing, and assessment instruments will be the same as in Phase I. This represents an opportunity to identify all potential responders to risperidone as an augmenting agent.

Safety Evaluations

* Baseline, week 4, and week 8 if applicable: Blood-cell-count (CBC) and differential, electrolytes, thyroid and kidney function tests, and urine pregnancy test.
* Vital signs and weight; baseline and weekly thereafter
* Side-effect questionnaire; baseline and weekly thereafter

Drug Accountability

A medication log will be maintained for each subject detailing dose and schedule on a daily basis. At each weekly visit subjects will be provided with enough medication for one-week of treatment plus an additional 2 days supply for safety. They will be required to return any unused medication at the end of each week. All drug supplies will be stored in a locked cabinet.

ELIGIBILITY:
Inclusion Criteria:

1. Boys and girls ages 7 to 12 years, inclusive
2. Medical/neurological clearance
3. Meets DSM-IV diagnosis of ADHD
4. Treatment with a stimulant medication during the last three weeks
5. Failure to respond to stimulant medication as documented by:

   1. Three acts of aggression in the past week, two of which must be acts of physical aggression against other people, objects, or self
   2. Aggression Questionnaire (AQ) Predatory-Affective index score of 0 or below. This indicates primarily an affective or impulsive subtype of aggression
   3. Minimum CGI scale rating of 4 (moderately ill)
6. IQ > 75 -

Exclusion Criteria:

1. Major medical problems such as cardiac, renal, thyroid diseases, and seizure disorder
2. History of alcohol or substance abuse within the last 4 weeks
3. Previous adequate treatment with risperidone (2 mg/day for at least 4 weeks)
4. Acutely suicidal or homicidal
5. Unable to sign informed consent

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25
Dates: Start 2003-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Children' Aggression Scale

SECONDARY OUTCOMES:
Clinical Global Impressions

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Armenteros, MD, Principal Investigator — Jorge L. Armenteros, M.D., P.A.
Locations (1):
- Jorge L. Armenteros, M.D., P.A., Coral Gables, Florida, United States